CLINICAL TRIAL: NCT05348421
Title: Comparing the Postoperative Analgesic Effect of Fascia Transversalis Plane Block Versus Pericapsular Nerve Group Block for Hip Surgery in Pediatrics: A Randomized Controlled Clinical Trial
Brief Title: Postoperative Analgesic Effect of Two Peripheral Nerve Blocks for Hip Surgery in Pediatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Ahmed Ismail Elnaggar, Principal Investigator, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB NO: 00012098, SN: 0305476
Record Dates: First submitted 2022-04-05; First posted 2022-04-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Pain, Postoperative; Developmental Dysplasia of the Hip; Regional Anesthesia Morbidity
Keywords: Fascia Transversalis plane block; pericapsular nerve group block; developmental dysplasia of the hip; postoperative analgesia; pediatric; hip surgery
MeSH Terms: conditions — Pain, Postoperative; Developmental Dysplasia of the Hip

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the ultrasound-guided fascia transversalis plane block (Experimental): The TFPB will be performed while the participant is in the supine position. a high-frequency linear ultrasound probe (5-13 MHz) will be placed transversely in the midaxillary line between the iliac crest and the costal margin. After the external oblique, internal oblique, transversus abdominis muscle, and quadratus lumborum (QL) muscle will be identified.
  Interventions: Procedure: FTPB
- The ultrasound guided Pericapsular Nerve Group block (Experimental): while the participant is in the supine position, a linear ultrasound probe will be initially placed in a transverse plane over the anterior inferior iliac spine (AIIS) and then aligned with the pubic ramus by rotating the probe counterclockwise approximately 45 degrees; In this view, the ilio-pubic eminence (IPE), the iliopsoas muscle and tendon, the femoral artery, and pectineus muscle will be observed.
  Interventions: Procedure: PENG Block

INTERVENTIONS:
Procedure: FTPB — A 22-gauge needle will be advanced from anterior using an in-plane technique and passed through the posterior 'tail' of the transversus muscle. the local anesthetic solution of 0.25% bupivacaine will be injected for a total volume of 0.5 ml/kg will be injected to separate the transversalis fascia from the transversus muscle.
  Other Names: Fascia Transversalis Plane Block
  Arms: the ultrasound-guided fascia transversalis plane block
Procedure: PENG Block — A 22-gauge, 80-mm needle will be inserted from lateral to medial in an in-plane approach to place the tip in the musculofascial plane between the psoas tendon anteriorly and the pubic ramus posteriorly where the local anesthetic solution of 0.25% bupivacaine will be injected for a total volume of 0.5 ml/kg
  Other Names: Pericapsular Nerve Group block
  Arms: The ultrasound guided Pericapsular Nerve Group block

SUMMARY:
Hip joint surgery for developmental dysplasia of the hip (DDH) in children is extremely painful and associated with considerable postoperative pain despite the use of systemic opioids. Caudal anesthesia and lumbar plexus block (LPB) were still the most common regional anesthesia techniques for perioperative analgesia in children undergoing this type of surgery. recently, pediatric anesthesiologists don't consider choosing both techniques because of potential complications such as intravascular and intrathecal injection, and urine retention. novel peripheral nerve blocks have been advocated in pediatrics to avoid the aforementioned complications such as PEricapsular Nerve Group (PENG) block, Quadratus Lumborum Block (QLB), and Fascia Transversalis Plane Block (FTPB) The objective of the current study is to assess the analgesic efficacy of ultrasound-guided FTPB versus ultrasound-guided PENG block in pediatric patients undergoing open hip surgery for DDH

DETAILED DESCRIPTION:
During the pre-anesthesia check-up visit, the proposed intervention will be discussed with the eligible participant's parents or caregivers including data about the aim, the advantages, and the expected side effects, and then a detailed written informed consent will be obtained before recruitment and randomization.

All participants will be premedicated with 0.5mg/kg oral midazolam about 30min before being admitted to the operating room. The routine standard monitoring including electrocardiography (ECG), non-invasive blood pressure (NIBP), pulse oximetry for blood oxygen saturation (SpO2), temperature probe, and end-tidal CO2 (EtCO2) will be applied to all participants. Induction of general anesthesia (GA) will be performed using a face mask with sevoflurane inhalation in oxygen starting with 2% up to 8% till complete loss of consciousness after that peripheral intravenous (IV) line will be secured where fentanyl 1 μg/kg and followed by cisatracurium 0.15mg/kg to facilitate orotracheal intubation. Anesthesia will be maintained by using isoflurane 1.2-1.5% in oxygen air mixture 50%:50% in addition to incremental cisatracurium 0.03mg/kg.

After induction of GA, the eligible participants will be randomly assigned to one of two equal groups either FTPB or PENG block.

In both interventional group participants, the assigned block will be performed after induction of GA by the same investigator who will have no further role in the study. Surgery will be started about 15 minutes after performing the block.

Fentanyl 1μg/ kg will be administrated intraoperatively in the case of inadequate analgesia which is defined as an increase of heart rate (HR) and/or mean arterial blood pressure (MAP) more than 20% above the pre-operative values. At the end of the surgery, isoflurane will be switched off and extubation will be done after reversal of muscle relaxant with neostigmine 0.05 mg/kg and atropine 0.02 mg/kg where the participants will be transferred to the Post-Anesthesia Care Unit (PACU). Paracetamol (15 mg/kg) will be administered IV every 6 hours in all participants.

ELIGIBILITY:
Inclusion Criteria:

* American society association (ASA) physical status class I - II.
* Participants who will be scheduled for an elective unilateral open hip surgery for correction of DDH under general anesthesia.

Exclusion Criteria:

* Participants with respiratory disease, renal or hepatic insufficiency.
* Infection of the skin in the puncture area.
* Coagulopathy.
* Allergy against any of the drugs to be used (bupivacaine).
* Neuromuscular disease.
* Obesity (body mass index, BMI >30).
* Bilateral hip surgery or previous hip surgery.
* Previous analgesic medication or chronic pain under treatment.
* previously known neurological pathologies or central nervous system disorders.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
The time until the first rescue analgesic requirement postoperatively | the first postoperative 48 hours
  Postoperative pain will be assessed by Face, leg, activity, cry, consolability (FLACC) score by the attending physician either in the PACU or in the surgical ward which ranges from a minimum score of zero (relaxed & comfortable) to a maximum of 10 (severe discomfort &pain). Morphine IV 0.1 mg/kg will be given as rescue analgesia if the FLACC score will be more than 3.

CONTACTS AND LOCATIONS:
Overall Officials: Hisham M Gamal Eldine, MD, Study Director — Alexandria University
Locations (1):
- Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ortiz-Neira CL, Paolucci EO, Donnon T. A meta-analysis of common risk factors associated with the diagnosis of developmental dysplasia of the hip in newborns. Eur J Radiol. 2012 Mar;81(3):e344-51. doi: 10.1016/j.ejrad.2011.11.003. Epub 2011 Nov 26. PMID 22119556
- [Background] Klisic PJ. Congenital dislocation of the hip--a misleading term: brief report. J Bone Joint Surg Br. 1989 Jan;71(1):136. doi: 10.1302/0301-620X.71B1.2914985. No abstract available.
- [Background] Gurkan Y, Aksu C, Kus A, Toker K, Solak M. One operator's experience of ultrasound guided lumbar plexus block for paediatric hip surgery. J Clin Monit Comput. 2017 Apr;31(2):331-336. doi: 10.1007/s10877-016-9869-x. Epub 2016 Mar 31. PMID 27033707
- [Background] Tsui BC, Berde CB. Caudal analgesia and anesthesia techniques in children. Curr Opin Anaesthesiol. 2005 Jun;18(3):283-8. doi: 10.1097/01.aco.0000169236.91185.5b. PMID 16534352
- [Background] Kao SC, Lin CS. Caudal Epidural Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:9217145. doi: 10.1155/2017/9217145. Epub 2017 Feb 26. PMID 28337460
- [Background] Suresh S, Chan VW. Ultrasound guided transversus abdominis plane block in infants, children and adolescents: a simple procedural guidance for their performance. Paediatr Anaesth. 2009 Apr;19(4):296-9. doi: 10.1111/j.1460-9592.2009.02958.x. PMID 19335342
- [Background] Chin KJ, McDonnell JG, Carvalho B, Sharkey A, Pawa A, Gadsden J. Essentials of Our Current Understanding: Abdominal Wall Blocks. Reg Anesth Pain Med. 2017 Mar/Apr;42(2):133-183. doi: 10.1097/AAP.0000000000000545. PMID 28085788
- [Background] Hebbard PD. Transversalis fascia plane block, a novel ultrasound-guided abdominal wall nerve block. Can J Anaesth. 2009 Aug;56(8):618-20. doi: 10.1007/s12630-009-9110-1. Epub 2009 Jun 4. No abstract available. PMID 19495909
- [Background] Serifsoy TE, Tulgar S, Selvi O, Senturk O, Ilter E, Peker BH, Ozer Z. Evaluation of ultrasound-guided transversalis fascia plane block for postoperative analgesia in cesarean section: A prospective, randomized, controlled clinical trial. J Clin Anesth. 2020 Feb;59:56-60. doi: 10.1016/j.jclinane.2019.06.025. Epub 2019 Jun 27. PMID 31255890
- [Background] Lopez-Gonzalez JM, Lopez-Alvarez S, Jimenez Gomez BM, Arean Gonzalez I, Illodo Miramontes G, Padin Barreiro L. Ultrasound-guided transversalis fascia plane block versus anterior transversus abdominis plane block in outpatient inguinal hernia repair. Rev Esp Anestesiol Reanim. 2016 Nov;63(9):498-504. doi: 10.1016/j.redar.2016.02.005. Epub 2016 Apr 8. English, Spanish. PMID 27067036
- [Background] Huang C, Zhang X, Dong C, Lian C, Li J, Yu L. Postoperative analgesic effects of the quadratus lumborum block III and transversalis fascia plane block in paediatric patients with developmental dysplasia of the hip undergoing open reduction surgeries: a double-blinded randomised controlled trial. BMJ Open. 2021 Feb 4;11(2):e038992. doi: 10.1136/bmjopen-2020-038992. PMID 33542037
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] Gerhardt M, Johnson K, Atkinson R, Snow B, Shaw C, Brown A, Vangsness CT Jr. Characterisation and classification of the neural anatomy in the human hip joint. Hip Int. 2012 Jan-Feb;22(1):75-81. doi: 10.5301/HIP.2012.9042. PMID 22344482
- [Background] Merkel SI, Voepel-Lewis T, Shayevitz JR, Malviya S. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs. 1997 May-Jun;23(3):293-7. PMID 9220806
- [Background] Charan J, Biswas T. How to calculate sample size for different study designs in medical research? Indian J Psychol Med. 2013 Apr;35(2):121-6. doi: 10.4103/0253-7176.116232. PMID 24049221
- [Background] Pannucci CJ, Wilkins EG. Identifying and avoiding bias in research. Plast Reconstr Surg. 2010 Aug;126(2):619-625. doi: 10.1097/PRS.0b013e3181de24bc. PMID 20679844
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343